CLINICAL TRIAL: NCT03556956
Title: Masitinib in Combination With FOLFIRI Versus Masitinib Alone, Versus Best Supportive Care, in Third or Fourth Line of Treatment of Patients With Metastatic Colorectal Cancer
Brief Title: Masitinib in Combination With FOLFIRI in Third or Fourth Line of Treatment of Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB12010
Record Dates: First submitted 2018-06-03; First posted 2018-06-14 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — masitinib

STUDY DESIGN:
Intervention Model Description: Prospective, multicentre, open-label, randomized, parallel groups, seamless phase 2-3 study to compare the efficacy and safety of masitinib in combination with FOLFIRI (irinotecan, 5-fluorouracil and folinic acid), versus Best Supportive Care in third or fourth line of treatment of patients with metastatic colorectal cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Masitinib plus FOLFIRI (Experimental): Masitinib in combination with FOLFIRI (irinotecan, 5-fluorouracil and folinic acid).
  Masitinib will be prescribed until disease progression (or treatment switch to next line of treatment), death, limiting toxicity or patient consent withdrawal.
  Interventions: Drug: Masitinib
- Best Supportive Care (No Intervention): Best Supportive Care (BSC) includes any concomitant medications or treatments: antibiotics, analgesics, radiation therapy for pain control (limited to bone metastases), corticosteroids, transfusions, psychotherapy, growth factors, palliative surgery, or any other symptomatic therapy necessary to provide BSC, except other investigational anti-tumor agents or anti-neoplastic chemo/hormonal/immuno-therapy.

INTERVENTIONS:
Drug: Masitinib — Tyrosine kinase inhibitor
  Other Names: AB1010
  Arms: Masitinib plus FOLFIRI

SUMMARY:
A prospective, multicentre, open-label, randomized, phase 2-3 study to compare the efficacy and safety of masitinib in combination with FOLFIRI (irinotecan, 5-fluorouracil and folinic acid) versus Best Supportive Care, in third or fourth line treatment of patients with metastatic colorectal cancer

DETAILED DESCRIPTION:
The objective is to compare the efficacy and safety of masitinib in combination with FOLFIRI (irinotecan, 5-fluorouracil and folinic acid) versus Best Supportive Care in third or fourth line treatment of patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non-resectable metastatic colorectal cancer with histological or cytological documentation of adenocarcinoma of the colon or rectum.
* Patient in third line or fourth line of treatment for metastatic colorectal cancer.
* Patient with measurable lesions according to RECIST criteria (version 1.1).
* Patient with ECOG equal to or less than 2.
* Patient with adequate organ function
* Other inclusion criteria may also apply

Exclusion Criteria:

* Prior treatment with masitinib, or any other tyrosine kinase inhibitor for the treatment of malignancy, except regorafenib.
* More than 3 prior chemotherapy regimens for metastatic colorectal cancer.
* Pregnant, intent to be pregnant, or nursing female patient
* Patient with any chronic inflammatory bowel disease
* Patient treated for a cancer other than colorectal cancer within five years before enrollment, with the exception of basal cell carcinoma or cervical cancer in situ.
* Other exclusion criteria may also apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | From day of randomization to death, assessed for a maximum of 60 months
  Overall survival (0S) is defined as time in months from the randomization date to the date of death due to any cause. If a patient is not known to have died, then OS will be censored at the date of last known date patient alive.

SECONDARY OUTCOMES:
Survival rates | Every 24 weeks, assessed up to 60 months
  Survival rate, defined as the proportion of patients alive at each time point, estimated with Kaplan-Meier distribution
Progression Free Survival (PFS) | From day of randomization to disease progression or death, whichever came first, assessed up to 60 months
  Progression Free Survival (PFS) is defined as the time from the randomization date until the date of earliest evidence of disease progression or death, for participants who progressed or died before subsequent cancer therapy. Disease progression will be assessed by the investigator on CT scan according to RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Taieb, MD, Principal Investigator — Hôpital Européen Georges Pompidou, Paris, France
Locations (5):
- University Hospital Olomouc, Olomouc, Czechia
- Chu - Hopitaux de Rouen, Rouen, France
- Omsk Clinical oncology dispensary, Omsk, Russia
- Hospital Madrid Norte San Chinarro, Madrid, Spain
- Hammersmith Hospital Imperial College Healthcare Nhs Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided